CLINICAL TRIAL: NCT02242669
Title: Enhancing Outcomes, Reducing Costs: Evaluating Peer Support for Mood Disorders
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, John F. Kelly, Associate Professor of Psychiatry Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2014P000153; R21MH101271-02 (NIH)
Record Dates: First submitted 2014-08-18; First posted 2014-09-17 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Depression; Bipolar Disorders; Mood Disorders
MeSH Terms: conditions — Depression; Bipolar Disorder; Mood Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- AIM 1: 200 current DBSA participants.
- AIM 2: 60 new DBSA attendees with mood disorders who have attended their first meeting in the past month.
- AIM 3: 100 matched control group individuals with mood disorders with no current or prior exposure to DBSA.

SUMMARY:
The purpose of this study to evaluate peer-led mutual help organizations (MHOs) that target individuals with psychiatric diagnoses such as mood disorders, and provide evidence either supporting the expansion of such groups and the development and testing of clinical procedures, or point toward reevaluation and development of alternative low-cost, community based approaches to promoting recovery among individuals suffering from these disorders.

DETAILED DESCRIPTION:
Participants will include up to 200 participants from The Depression and Bipolar Support Alliance (DBSA) for Aim 1. Aim 1 will measure characteristics of current DBSA members through cross-sectional surveys of demographics, clinical use history, and involvement in DBSA. 60 new DBSA members who began attending in the past month will be enrolled for Aim 2. Aim 3 will consist of 100 matched controls of people who have never attended a DBSA meeting. Assessments will be completed at McLean Hospital, in which a study staff member will thoroughly explain the study to participants. If participants are eligible for Aim 2, study staff will receive written consent from the participant.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1:
* 18 years of age or older
* Self-report a diagnosis of any type of mood disorder
* Attend DBSA meetings
* Aim 2:
* 18 years of age or older
* Self-report a diagnosis of any type of mood disorder
* Have attended their first meeting in the past month
* Aim 3:
* 18 years of age or older
* Self-report a diagnosis of any type of mood disorder
* Have never attended a DBSA meeting

Exclusion Criteria:

* Aim 1:
* Do not report a diagnosis of any type of mood disorder
* Have not attended a DBSA meeting
* Aim 2:
* Do not report a diagnosis of any type of mood disorder
* Have not attended a DBSA meeting
* Have attended their first meeting prior to a month before their assessment
* Aim 3:
* Do not report a diagnosis of any type of mood disorder
* Have attended a DBSA meeting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit participants from a large DBSA chapter at McLean Hospital. Subjects will be recruited at the beginning of the weekly meetings, through flyers, the DBSA website, and word of mouth. 200 current DBSA members and 60 new DBSA members will be assessed for Aims 1 and 2, respectively. 100 people who have never attended a DBSA will be assessed for Aim 3 and will be recruited from MGH and McLean Hospitals through the use of flyers, clinic announcements, and via our online clinical and research infrastructures. Participants in all Aims must be 18 years or older and self-report a diagnosis of any type of mood disorder. For Aims 1 and 2, participants must have attended at least one DBSA meeting.
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2014-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Systematically gather empirical estimates of the characteristics of current DBSA participants through a cross-sectional survey of demographics, clinical service, and past and current DBSA attendance, involvement, and subjective benefits. | Up to 24 months
  The goal is to describe and characterize DBSA participants and obtain information on subjective benefits.
Provide estimates of rates of attendance, retention in, and discontinuation from DBSA for new DBSA members with mood disorders. | Up to 24 months
  Determine which DBSA participants are more likely to attend more frequently/become more engaged.
Conduct a prospective between-group investigation comparing new DBSA members to a matched control group with no prior exposure to DBSA in order to test for beneficial affects of DBSA over a 6-month follow up. | Up to 24 months
  Compare new DBSA members to a matched control group in order to test for any potential incremental beneficial effects from DBSA participation.

CONTACTS AND LOCATIONS:
Overall Officials: John F Kelly, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts